CLINICAL TRIAL: NCT05343858
Title: Pilot Study to Evaluate the Effect of the Consumption of Two Unicellular Microalgae (Chlorella Vulgaris and Arthrospira Platensis (Spirulina)) on Metabolic Syndrome Biomarkers in Overweight / Obese Subjects With Altered Lipid Profile
Brief Title: Pilot Study to Evaluate the Effect of Two Microalgae Consumption on Metabolic Syndrome
Acronym: ALGAENERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: AlgaEnergy, S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HULP 5296
Record Dates: First submitted 2019-09-06; First posted 2022-04-25 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Syndrome
Keywords: microalgae; lipid profile; metabolic syndrome; pilot
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Spirulina platensis (Experimental): 10 volunteers will consume 16g / day (in 2 doses of 8g) of a nutritional supplement of Spirulina platensis
  Interventions: Dietary Supplement: Experimental: Group 1: Spirulina platensis
- Group 2: Chlorella vulgaris (Experimental): 10 volunteers will consume 16g / day (in 2 doses of 8g) of a nutritional supplement of Chlorella vulgaris
  Interventions: Dietary Supplement: Experimental: Group 2: Chlorella vulgaris
- Group 3: Control (Placebo Comparator): 10 volunteers will consume 16g / day (in 2 doses of 8g) of a control supplement
  Interventions: Dietary Supplement: Placebo Comparator: Group 3: Control

INTERVENTIONS:
Dietary Supplement: Experimental: Group 1: Spirulina platensis — 16 g/day (two doses of 8g)
  Arms: Group 1: Spirulina platensis
Dietary Supplement: Experimental: Group 2: Chlorella vulgaris — 16 g/day (two doses of 8g)
  Arms: Group 2: Chlorella vulgaris
Dietary Supplement: Placebo Comparator: Group 3: Control — 16 g/day (two doses of 8g)
  Arms: Group 3: Control

SUMMARY:
The purpose of this study is to evaluate the effect of the consumption of two microalgae Chlorella vulgaris and Arthrospira platensis (Spirulina) on some biomarkers of metabolic syndrome: Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, Apolipoprotein A and Apolipoprotein B, in overweight / obese subjects with altered lipid profile.

DETAILED DESCRIPTION:
A randomized, parallel, and double-blind pilot study with 3 study arms is being performed to evaluate the effect of the consumption of two unicellular microalgae: Chlorella vulgaris and Arthrospira platensis (Spirulina).

The investigators included 30 participants between 18 and 65 years (BMI ≥25 and <40 kg / m2). All volunteers will be randomized into 3 study groups, and participants will receive the 3 different study products during 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years old.
* Body Mass Index (BMI) ≥25 and <40 kg/m2.
* Cardiovascular risk <10%
* Adequate cultural level and understanding
* Agree to participate in the study

Exclusion Criteria:

* Subjects with BMI ≥40 or <25 kg /m2
* Subjects diagnosed with Diabetes Mellitus.
* Subjects with dyslipidemia on pharmacological treatment
* Subjects with hypertension on pharmacological treatment
* Subjects with established diagnosis of eating disorder
* Smokers or those subjects with high alcohol consumption
* Subjects under pharmacological treatment
* Subjects with large weight fluctuations of more than 4 kg or who have undergone in six months a weight loss diet
* Subjects with sensory problems
* Subjects with gastrointestinal diseases that affect the digestion or absorption of nutrients
* Pregnant or breastfeeding women
* Women with menstrual irregularities
* Subjects with intense physical activity
* Subjects with food allergies to meals included in breakfast, study product or lunch or that reject their consumption
* Subjects with a diagnosis of celiac disease or a gluten intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Serum cholesterol | Change from baseline at 30 days
  Biomarker of metabolic syndrome
Serum HDL | Change from baseline at 30 days
  Biomarker of lipid profile quality
Serum LDL syndrome biomarker | Change from baseline at 30 days
  Biomarker of lipid profile quality
Triglycerides (TAG) | Change from baseline at 30 days
  Biomarker of lipid profile quality
Apolipoprotein A | Change from baseline at 30 days
  Metabolic syndrome biomarker
Apolipoprotein B | Change from baseline at 30 days
  Metabolic syndrome biomarker

SECONDARY OUTCOMES:
Blood count | Change from baseline at 30 days
  Concentration of blood
Body weight | Change from baseline at 30 days
  Changes on anthropometric characteristics
Tolerance | Change from baseline at 30 days
  Occurrence and frequency of gastrointestinal symptoms
Body Mass Index | Change from baseline at 30 days
  Changes on anthropometric characteristics
Waist circumference | Change from baseline at 30 days
  Changes on anthropometric characteristics
Adherence | Change from baseline at 30 days
  Changes in the number of consumed pills
Sensory perception Visual Analog Scale (VAS) rate from 1 to 100 related with flavor, aro | Change from baseline at 30 days
  Visual Analog Scales (VAS) with a range between 0 (negative score) and 10 (positive score) related to taste, smell, texture, satiety and fullness
Dietary intake | Change from baseline at 30 days
  Changes in diet composition through 24-hour dietary record
Glucose | Change from baseline at 30 days
  Concentration of glucose
Urate | Change from baseline at 30 days
  Concentration of safety marker
Creatinine | Change from baseline at 30 days
  Concentration of creatinine
Calcium | Change from baseline at 30 days
  Concentration of minerals

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez-Candela, Principal Investigator — La Paz University Hospital
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain